CLINICAL TRIAL: NCT04335110
Title: Assessing Acceptability, Cost, and Efficacy of STELLA-Support Via Technology: Living and Learning With Advancing AD
Brief Title: Assessing Acceptability, Cost, and Efficacy of STELLA-Support Via Technology
Acronym: STELLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Walter Dawson, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00019306; 2P30AG024978-16 (NIH)
Record Dates: First submitted 2020-03-11; First posted 2020-04-06 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Dementia; Alzheimer Disease; Caregiver Burnout; Family Members
MeSH Terms: conditions — Dementia; Alzheimer Disease; Caregiver Burden | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Care Partners and Persons with Dementia. Up to 40 Care Partners and their 40 care-recipients with ADRD will participate in this study. The primary focus of this study is on Care Partners, however, we will gather subjective and objective data on participants with Alzheimer's Disease and Related Dementias (ADRD) to assess the effect of the intervention on Care Partner affective responses to caregiving and quality of life for both. STELLA participants will be recruited from the existing cohort of patients, and their Care Partners, who are enrolled in the Oregon Roybal Center for CAre Support Translational Research Advantaged by Integrating Technology) ORCASTRAIT Life Laboratory (OSLL).
  Interventions: Behavioral: STELLA (Support via TEchnology: Living and Learning with Advancing Alzheimer's disease and related dementias)

INTERVENTIONS:
Behavioral: STELLA (Support via TEchnology: Living and Learning with Advancing Alzheimer's disease and related dementias) — STELLA consists of 8 sessions: 4 sessions one-to-one, with the Care Partner and a Guide, and then 4 sessions with one Guide with up to four Care Partners (total small group will include as few as two and as many as 4 Care Partners) Each weekly session takes about 1 hour. The first four sessions allow for development of the Care Partner-Guide working relationship. In these sessions, the Care Partners identify behaviors (both the person with dementia's and the Care Partner's) which are upsetting to the family. Care Partners will be taught to use an Activator, Behavior, Consequence (ABC) approach to identify activators of behaviors, the behaviors, and consequences of the behaviors. After they identify the ABCs, they will develop a plan to address the behavior and then test it. After the four one-to-one sessions, Care Partners will meet in small groups with a Guide. Effective communication strategies, engagement in pleasant events, and coping will be addressed.

SUMMARY:
STELLA (Support via Technology Living and Learning with Advancing Alzheimer's disease and related dementias) is a multicomponent video-conference based intervention that aims to help family members caring for persons of dementia as well the person with dementia. The goal of this intervention is to reduce upsetting behaviors and care partner burden. Caring for a family member with Alzheimer's disease or related dementia (ADRD) can come with many burdens that affect not only the care partners' physical and psychological health but also barriers to access. Due to factors such as distance and cost, Internet-based interventions like STELLA are a great alternative to in-person interventions because it can still address the specific needs of families living with dementia. The hypothesis of this study is that care partners will show significant improvements in burden and depression following the intervention. STELLA is also designed to facilitate effective management of behavioral and psychological symptoms of dementia (BPSD). To accomplish this, up to 40 care partners and their 40 care recipients with Alzheimer's disease and related dementias will participate in an 8-week intervention with the support of a Guide (e.g. nurse or social worker). However, the primary focus of this study is on care partners. With the support of a Guide, care partners will identify strategies to address upsetting behaviors in the moderate to late stages of dementia. More specifically, a Guide will help care partners identify and modify distressing behavioral symptoms of dementia. Based on quantitative and qualitative approaches, the effect of the intervention on care partner affective symptoms, including depression and burden, as well as quality of life for both the care partner and the person with dementia will be assessed.

DETAILED DESCRIPTION:
Introduction and Specific Aims:

Family members who care for those with Alzheimer's disease and related dementias (ADRD) may find a sense of meaning, opportunity and power in their evolving role, but they may also find the experience burdensome, leading to depression, anxiety and grief. Caregiving can also have negative effects on health, including impairments in cardiovascular health, immune function, restorative sleep and cognitive function. As care demands build over the long duration of disease, the quality of life for the care dyad (the person with dementia, (PwD) and their care partner (CP)) is affected and the risk of placement for the PwD increases. Interventions that reduce the CP affective and physical burden, and delay PwD placement are available to support the 16 million ADRD CPs in the United States, but access to them is limited by a number of factors, including geographic distance, financial resources and stigma.

Internet-based videoconferencing technology (also known as "telehealth") is making education and support interventions more accessible for families living with ADRD. These interventions have had small to moderate effects on reducing CP burden and depression and good consumer acceptance. However, despite evidence that CPs prefer individualized interventions with real-time counselors, most telehealth interventions are group-based, automated and not tailored to stages of disease. Also, while the telehealth interventions target important aspects of the CP affective experience (burden, depression), few address sleep issues or the cognitive dysfunction that can result from caregiving. Further, limited information is available about the mechanisms of action of these technology-based interventions.

To address the need for personalized, real-time educational interventions for families caring for those in moderate to late-stage dementia, we designed Tele-STELLA (Support via TEchnology: Living and Learning with ADRD). Tele-STELLA uses videoconferencing to connect nurse consultants with CPs, in both one-to-one and then small group sessions. STELLA uses cognitive behavioral techniques to guide CPs in strategies to reduce the emotional, cognitive and physical effects of upsetting behavioral symptoms of dementia. Pilot testing of STELLA prototypes found that the intervention reduced burden. Focus groups revealed that CPs liked the one-to-one telehealth format, but did not like the abrupt cessation after completing the 8 weekly sessions. They asked for opportunities to connect with other caregivers to sustain support.

There are few known telehealth interventions that use combined one-to-one and group sessions. This novel study, co-developed with CPs, will provide feasibility and efficacy data and help understand the mechanisms of change for this intervention. Further, this study will be one of the first to use objective data from the ORCASTRAIT LL to learn about Tele-STELLA's mechanisms of behavior change.

Phase 1 assesses the STELLA intervention, Phase 2 assesses costs and the effect of the intervention on costs.

Phase 1

1. Using quantitative and qualitative approaches, assess feasibility and participant acceptability of (a) STELLA, and (b) the assessment methods (subjective measures and unobtrusive objective monitoring).
2. Using quantitative strategies, assess the preliminary effect of STELLA on (a) the affective impact of caregiving, Care Partner cognitive function and person with dementia quality of life, and on (b) Care Partner and person with dementia objective digital behavioral biomarkers (activity, sleep and time together).
3. Test the feasibility of employing digital behavioral biomarker data, combined with qualitative Care Partner feedback, to assess mechanisms of behavior change before, during and after the STELLA intervention.

Phase 2

1. Quantify the costs of delivering the STELLA intervention.
2. Quantify the cost efficacy of STELLA in relation to BPSD frequency and CP reactivity and assess the relationship between costs, BPSD, and care partner burden.

H1: There is a relationship between BPSD and cost: More BPSD behaviors and more CP reactivity to the BPSD are associated with higher out-of-pocket and implicit costs for families living with dementia.

H2: There is a relationship between out-of-pocket and implicit costs and objective measures of burden identified in the ORCASTRAIT Living Lab continuous home assessment. Higher objective burden will correlate with higher implicit and out-of-pocket costs.

STELLA is an ancillary study embedded in the Oregon Roybal Center for CAre Support Translational Research Advantaged by Integrating Technology (ORCASTRAIT) parent study (IRB#20236).

THEORETICAL FRAMEWORK AND MECHANISMS OF ACTION: Tele-STELLA is framed by Vitaliano et al's model which hypothesizes that CP stress exposure catalyzes a cascade of concerns, including psychological, physiological and cognitive strain. The original model places the caregiver at the top of the model as the recipient of a stressor. However, the PwD also experiences stressors, such as CP disengagement. Thus, we include the PwD, who is also vulnerable to the stress of caregiving, at the top of the model. By addressing behavioral symptoms in both the CP and the PwD, it is hypothesized that Tele-STELLA will be feasible and acceptable to families, will reduce the negative effects of ADRD on the family, and that objective feedback (provided by digital biomarker data) will inform the efficacy of the intervention and the mechanisms of behavior change.

Significance Providing care for a family member with Alzheimer's disease or a related dementia (ADRD) is both rewarding and risky. CPs exposed to chronic stress, often over years, are susceptible to physical and psychological ailments. In addition, the caregiving experience increases the risk of cognitive impairment in CPs, with spousal CPs being particularly vulnerable, thus potentially perpetuating a cycle when yet another family member has to care for the former CP. Effective interventions that reduce caregiver burden and reduce health risks are available, but various factors impede CP participation, including distance, cost, behavioral symptoms of dementia, stigma and social anxiety. Recognizing the need to reduce barriers to access, scientists have turned to Internet-based interventions. Recent research indicates that multi-component technology-facilitated interventions which allow CP engagement with health professionals are effective and favored by caregivers. However, only a minority of studies allow for health professional engagement, and of these, only a handful provide real-time interaction. Hopwood et al concluded that, despite the fact that family needs vary across ADRD stages, the interventions reviewed were not targeted to a specific stage of ADRD.

We have completed two pilot studies using Internet-based CP interventions. These studies tested the feasibility and consumer acceptability of the evidence-based, Staff Training in Assisted-living Residences - Caregivers (STAR-C) intervention, the precursor to Tele-STELLA, when delivered via telehealth. Qualitative data revealed the telehealth intervention was acceptable to CPs and preferred over a potential in-home ("live") intervention. We found that burden was reduced, but depression was not. This may be because the interaction with the nurse consultant formally ended with the concluding Session 8, leaving CPs with a sense of isolation, as this CP commented: "I went through withdrawals… I wanted to call her (the nurse consultant)-who can I turn to?" The prototype interventions did not include meaningful opportunities for CPs to interact with each other post-intervention. CPs felt their support vanished and did not like "the fact that it was over". Participants advised that future interventions should include both one-to-one sessions and one-to-multiple sessions.

Based on the qualitative and quantitative data from the pilot work Tele-STELLA was designed to address the specific needs of families living with dementia. Tele-STELLA is a multi-component, tailored intervention that begins with one-to-one sessions with each CP and nurse consultant, then links CPs to each other in a meaningful way to sustain support post intervention. Tele-STELLA is designed for families living in the later stages of dementia, where behavioral symptoms are more prominent and distressing for all.

Innovation This pilot is innovative in several ways. First, we are testing a new intervention format (blended one-to-one and one-to three) using an online environment (Internet-based videoconferencing technology). Second, we are examining novel strategies for assessing the effect of the intervention and mechanisms of action using unobtrusive, objective monitoring of digital behavioral biomarkers (sleep, time together, activity). Finally, we are collecting data (saved video and audio files) that can be used for future objective assessment of dyad well-being, such as assessing conversational dynamics through linguistic analysis of session interactions or employing facial recognition techniques to assess CP emotions. Taken together, this pilot will set the stage to advance caregiving science beyond traditional, earthbound approaches.

ELIGIBILITY:
Care Recipient Inclusion:

* Diagnosis of Alzheimer's Disease and Related Dementias (ADRD), moderate to late stages
* Exhibits 2 or more behaviors listed on Revised Memory and Behavioral Problems (RMBP) that are bothersome to the Care Partner and occur 3 or more times/week at study enrollment
* Family member of Care Partner (this can be a relative, spouse or close kin that is considered family)

Care Recipient Exclusion:

* Dementia not related to ADRD
* Unable to leave Care Partner during Care Partner training
* Early stage dementia, as defined by a Montreal Cognitive Assessment (MoCA) of about 15/30 or higher.

Care Partner Inclusion:

* Adult caring for family member with ADRD
* Lives with care recipient OR spends at least 4 hours/week with care recipient
* Age of 18 years or older
* Speak English
* Own a computer/device with a reliable internet connection and compatible operating system

Care Partner Exclusion:

* Unable to find activity for care recipient during training which would allow Care Partner to work privately, one-on-one during training
* Completed similar telehealth intervention within the last year
* Hearing and vision problems severe enough to prevent participation
* Unwilling or unable to adequately follow study instructions and participate in study procedures

Inclusion for Care Recipient and Care Partner:

Participate in Oregon Roybal Center for CAre Support Translational Research Advantaged by Integrating Technology (ORCASTRAIT) (IRB#20236) Participant in the ORCASTRAIT study (IRB # 20236)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Dawson, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Layton Aging and Alzheimer's Disease Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available upon request to our Alzheimer's Disease Research Center.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 1/2021, available indefinitely
Access Criteria: Requests need to made to the PI at the Oregon Alzheimer's Disease Research Center (OARDC). A short data request form will need to be submitted to the OADRC

REFERENCES:
- [Derived] Dawson WD, Mattek N, Gothard S, Kaye J, Lindauer A. Ascertaining Out-of-Pocket Costs of Dementia Care: Feasibility Study of a Web-Based Weekly Survey. JMIR Form Res. 2024 Sep 25;8:e56878. doi: 10.2196/56878. PMID 39321453

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Administrative delays and COVID interference caused substantial delays in enrollment. Further enrollment required initial enrollment in the parent study, thus limiting recruitment pool. Recruitment started in Winter 2021, ending in Spring 2022.
Pre-assignment Details: Participants were assigned to care partner group (intervention) or care recipient (no intervention). The majority of participants that were referred to STELLA from ORCASTRAIT were eligible for the study.
Groups:
- Intervention: STELLA participants were be recruited from the existing cohort of patients who were enrolled in the Oregon Roybal Center for CAre Support Translational Research Advantaged by Integrating Technology) ORCASTRAIT Life Laboratory (OSLL).
  STELLA (Support via TEchnology: Living and Learning with Advancing Alzheimer's disease and related dementias): STELLA consists of 8 sessions: 4 sessions one-to-one, with the Care Partner and a Guide, and then 4 sessions with one Guide with up to four Care Partners (total small group will include as few as two and as many as 4 Care Partners) Each weekly session takes about 1 hour. The first four sessions allow for development of the Care Partner-Guide working relationship. In these sessions, the Care Partners identify behaviors (both the person with dementia's and the Care Partner's) which are upsetting to the family. Care Partners will be taught to use an Activator, Behavior, Consequence (ABC) approach to identify activators of behaviors, the behaviors, and consequences of the behaviors. After they identify the ABCs, they will develop a plan to address the behavior and then test it. After the four one-to-one sessions, Care Partners will meet in small groups with a Guide. Effective communication strategies, engagement in pleasant events, and coping will be addressed.
- Care Recipient: Care recipients did not receive the intervention
Period: Overall Study
Arm/Group | Intervention | Care Recipient
Started (Care partners were enrolled in Spring of 2021, completing in Spring 2023) | 14 | 14
Completed | 13 | 12
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Fourteen care partners and 14 care recipients enrolled
Groups:
- Intervention: Care Partners for persons with dementia
- Care Recipients: Care recipients
- Total: Total of all reporting groups
Arm/Group | Intervention | Care Recipients | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: separate values for care partners and care recipients
  years
    number analyzed (Participants) | 13 | 13 | 26
    (all) | 72 (8) | 76.6 (9.8) | 74.4 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — race of participants Population: no underrepresented individuals
  Participants
    number analyzed (Participants) | 13 | 13 | 26
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 13 | 13 | 26
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Revised Memory and Behavior Problems Checklist
Description: Care recipient frequency of behaviors and caregiver reactions to behavioral symptoms. The scale measures how often a behavior occurs (Frequency, "F") and how much the caregiver reacts to it (Reactivity, "R"). Range for both scales is 0-96, lower scores are better. Subscales are not combined.
Time Frame: The RMBPC is assessed 1 week prior to the 8-week intervention (pre), then 1 week after the intervention (post)
Population: Pre/post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: Caregivers for family members with dementia
- Care Recipients: Persons with dementia
Arm/Group | Intervention | Care Recipients
Number analyzed (Participants) | 13 | 13
units on a scale
  RMPBC, F Pre | NA (NA) — The Frequency Scale on the RMBPC is the # of behaviors for the person with dementia and does not apply to the caregivers | 41.5 (12)
  RMBPC, F, Post RMBPC, F, post | NA (NA) — The Frequency Scale on the RMBPC is the # of behaviors for the person with dementia and does not apply to the caregivers | 39.5 (13.9)
  RMBPC, R, Pre | 27.5 (14.9) | NA (NA) — The Reactivity Scale on the RMBPC is the caregiver's reaction to the behaviors and does not apply to the care recipients
  RMBPC, R, Post | 24.7 (13) | NA (NA) — The Reactivity Scale on the RMBPC is the caregiver's reaction to the behaviors and does not apply to the care recipients

2. Primary Outcome: Center for Epidemiological Studies Depression Scale
Description: Caregiver depression symptoms, Range 0-30, lower scores indicate less depression (better). Depression is only measured for the caregivers, not the care recipients with dementia (only 1 group)
Time Frame: 1 week prior to the 8-week intervention (pre), then 1 week after the intervention (post)
Population: 1 week prior to the 8-week intervention (pre), then 1 week after the intervention (post)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- One Arm Only (Caregivers): Caregivers
Arm/Group | One Arm Only (Caregivers)
Number analyzed (Participants) | 13
units on a scale
  CESD Pre | 9.9 (7.2)
  CESD Post | 9.5 (6.7)

3. Secondary Outcome: Desire to Institutionalize (DTI) Scale
Description: Care partner intention to place person with dementia in care facility. This only applies to caregivers.
Time Frame: Measured at study entry only
Population: Assesses caregivers desire to place person with dementia
Measure: Count of Participants; unit: Participants
Groups:
- Desire to Institutionalize: DTI is for caregivers only (not the persons with dementia).
Arm/Group | Desire to Institutionalize
Number analyzed (Participants) | 13
Participants
  Not likely | 11
  Possibly | 1
  very Likely | 1

4. Secondary Outcome: Marwit Meuser Caregiver Grief Index
Description: Caregiver anticipatory grief. Range is 0-90. Higher scores indicate worse grief. This only applies to the caregivers.
Time Frame: 1 week prior to the 8-week intervention (pre), then 1 week after the intervention (post)
Population: The MMCGI is only for caregivers (one group). This scale was not used with persons with dementia.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MMCGI Pre: MMCGI pre
Arm/Group | MMCGI Pre
Number analyzed (Participants) | 13
units on a scale
  Pre intervention | 60.9 (14.5)
  Post intervention | 58.9 (12.6)

5. Secondary Outcome: Feasibility and Participant Acceptability
Description: Measures how much participants find the intervention acceptable and feasible. This only applies to caregivers.
Time Frame: Measured only once by caregivers 1 week after 8-week intervention
Population: This is only for the caregivers (one group)
Measure: Number; unit: participants
Groups:
- Experience Survey: Information only
Arm/Group | Experience Survey
Number analyzed (Participants) | 13
participants
  It was easy for me to attend STELLA Visits | 12
  I could talk with the STELLA Guide easily and openly | 13
  I feel confident that I can use STELLA skills ot manage upsetting behaviors | 13
  I felt my privacy was respected during the STELLA visits | 13
  I felt comfortable discussing sensitive topics with my Guide | 13
  Comfortable talking with other participants | 13
  Easy to find activity for Care recipient | 11
  Good Technical support | 13
  Could see and hear others | 12
  Easy to connect | 12
  Liked working with other CPs | 13
  Prefer 1:1 for 8 weeks (no group) | 1
  Prefer group | 2
  Current format | 10
  Prefer in-person | 5
  Prefer video format | 8

6. Secondary Outcome: Quality of Life in Alzheimer's Disease (QOL-AD) Scale
Description: Quality of life for participants, both for caregivers and persons with dementia. The measure consists of 13 items, rated on a four point scale, with 1 being poor and 4 being excellent. Total scores range from 13 to 52, higher scores are better
Time Frame: 1 week prior to the 8-week intervention (pre), then 1 week after the intervention (post)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Caregivers: Family members caring for someone with dementia
- Care Recipients: Care recipients with dementia
Arm/Group | Caregivers | Care Recipients
Number analyzed (Participants) | 13 | 13
units on a scale
  QoL Pre | 37.1 (5.3) | 33.3 (7.7)
  QoL Post | 35.5 (6.2) | 34 (7.8)

7. Secondary Outcome: Sleep Duration
Description: Digital behavioral biomarker for effective impact of care on care partner sleep. Measured via electronic sleep mat
Time Frame: Measures sleep from enrollment to study end. Mean sleep hours one week prior to intervention (pre) and one week after intervention (post). Measured in hours (units on a scale)
Population: sleep duration
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Care Partners: hours of sleep with Emfit bed mat
- Care Recipients: care recipient emfit data
Arm/Group | Care Partners | Care Recipients
Number analyzed (Participants) | 12 | 12
hours
  pre intervention | 7.9 (1.5) | 8.9 (1.8)
  post intervention: number analyzed (Participants) | 12 | 8
  post intervention | 7.8 (1.8) | 9.2 (1.3)

ADVERSE EVENTS:
Time Frame: Duration of study participation (about 1.3 years)
Description: All caregivers are at low risk for adverse events. They are not "patients" and this is not a study that involves medication.
  Persons with dementia may have "adverse events" due to their advanced age and dementia status. However, these events are "expected" and not related to the study.
Groups:
- Intervention: Caregivers who participated in intervention
- Care Recipients: Care recipients (did not participate in intervention)
Arm/Group | Intervention | Care Recipients
All-Cause Mortality (participants affected / at risk) | 0/14 | 3/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 3/14
Other Adverse Events (participants affected / at risk) | 6/14 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=14) | Care Recipients (N=14)
Death (Nervous system disorders) | 0 (0) | 1 (1) — Not related to intevention
Death (Nervous system disorders) | 0 (0) | 1 (1) — Not related to intervention
Hospitalizaton: Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Covid and other URIs
Hospitalization GI (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hospitalization: Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=14) | Care Recipients (N=3)
care partner burden (Psychiatric disorders) | 2 (2) | 0 (0)
COVID (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Fall (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT04335110/Prot_SAP_001.pdf